CLINICAL TRIAL: NCT04468568
Title: Assessment of Maternal Blood Gas Changes When Using Atosiban and Terbutaline as Tocolytic Agents, During in Utero Repair of Myelomeningocele
Brief Title: In Utero Repair of Myelomeningocele: Atosiban Versus Terbutaline
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, Attending Anesthetist, University of Sao Paulo General Hospital
Other Study IDs: 00607219.4.0030.0099
Record Dates: First submitted 2020-03-01; First posted 2020-07-13 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Myelomeningocele; Terbutaline Adverse Reaction; Pregnancy; Malformation Central Nervous System
MeSH Terms: conditions — Meningomyelocele | interventions — atosiban; Terbutaline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atosiban: Intravenous Atosiban as main tocolytic agent
  Interventions: Drug: Atosiban
- Terbutaline: Intravenous Terbutaline as main tocolytic agent
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Atosiban — Atosiban intravenous. Dose: attack of 6.75 mg, and maintenance of 300 mcg / min for 3 hours, and 100 mcg / min for 21 hours.
  Groups: Atosiban
Drug: Terbutaline — Terbutaline intravenous. Dose: 2.5 mg in 500 mL saline, infusion rate of 30 mL / hr (150 mcg / h) during the surgery and for 24 hours.
  Groups: Terbutaline

SUMMARY:
Myelomeningocele is a malformation with high incidence, and it consists in a neural tube defect. Fetal intrauterine surgery is an alternative for correction, and it improves the prognosis of the fetus, but has an increased risk of maternal complications and premature labor, as it can occur due to uterine stimulation. It is therefore essential that tocolysis is performed before, during and after surgery, and the most commonly used tocolytics are terbutaline and atosiban. Terbutaline has no specificity and may have several adverse effects such as maternal acidosis.

DETAILED DESCRIPTION:
The objective of the study was to evaluate maternal blood gas alterations among cases that used atosiban tocolytic agent and cases with terbutaline in in utero repair of myelomeningocele. It consists of a retrospective cohort study. It included 25 patients, who were divided into two groups, depending on which agent they received as main tocolytic agent during the intrauterine fetal myelomeningocele repair: terbutalineor atosiban. The primary outcome was maternal arterial pH at the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years
* Single fetus pregnancy
* Fetus with myelomeningocele
* Gestational age from 19 to 26
* Fetus with normal karyotype

Exclusion Criteria:

* Multiple pregnancy
* Fetal abnormality not related to myelomeningocele
* Kyphosis greater than or equal to 30 degrees
* Placenta previa
* Maternal disease that increases the risk of pregnancy (insulin-dependent DM, hypertension poorly controlled)
* History of incompetent cervix
* Carrier of HIV, hepatitis B or hepatitis C
* Maternal-fetal isoimmunization
* Uterine Alteration
* Obesity (IMC greater than 30)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who underwent intrauterine myelomeningocele surgical repair in a tertiary obstetrical center (Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo), from November of 2017 to January of 2020.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Maternal arterial blood pH at the start of surgery | Right after intubation
  Arterial blood pH
Maternal arterial blood pH at the end of surgery | Before extubation
  Arterial blood pH
Maternal arterial blood pH at 120 minutes after surgery | Two hours after the end of surgery
  Arterial blood pH

SECONDARY OUTCOMES:
Short-term fetal repercussions | In the end of the surgery, before extubation
  Fetal heart rate in the immediate postoperative period
Long-term fetal repercussions | At the birth
  Gestational age at birth

CONTACTS AND LOCATIONS:
Overall Officials: Elaine I Moura, MD, Principal Investigator — Hospital das Clinicas; Hermann S Fernandes, PhD, Principal Investigator — Hospital das Clinicas
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan includes informations about the demographic sample, the results of the study and the statistical analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From October/2017 until January/2021
Access Criteria: Contact through email

REFERENCES:
- [Result] Ferschl M, Ball R, Lee H, Rollins MD. Anesthesia for in utero repair of myelomeningocele. Anesthesiology. 2013 May;118(5):1211-23. doi: 10.1097/ALN.0b013e31828ea597. PMID 23508219
- [Result] Boulet SL, Yang Q, Mai C, Kirby RS, Collins JS, Robbins JM, Meyer R, Canfield MA, Mulinare J; National Birth Defects Prevention Network. Trends in the postfortification prevalence of spina bifida and anencephaly in the United States. Birth Defects Res A Clin Mol Teratol. 2008 Jul;82(7):527-32. doi: 10.1002/bdra.20468. PMID 18481813
- [Result] Fichter MA, Dornseifer U, Henke J, Schneider KT, Kovacs L, Biemer E, Bruner J, Adzick NS, Harrison MR, Papadopulos NA. Fetal spina bifida repair--current trends and prospects of intrauterine neurosurgery. Fetal Diagn Ther. 2008;23(4):271-86. doi: 10.1159/000123614. Epub 2008 Apr 14. PMID 18417993
- [Result] Adzick NS, Thom EA, Spong CY, Brock JW 3rd, Burrows PK, Johnson MP, Howell LJ, Farrell JA, Dabrowiak ME, Sutton LN, Gupta N, Tulipan NB, D'Alton ME, Farmer DL; MOMS Investigators. A randomized trial of prenatal versus postnatal repair of myelomeningocele. N Engl J Med. 2011 Mar 17;364(11):993-1004. doi: 10.1056/NEJMoa1014379. Epub 2011 Feb 9. PMID 21306277
- [Result] Fisk NM, Gitau R, Teixeira JM, Giannakoulopoulos X, Cameron AD, Glover VA. Effect of direct fetal opioid analgesia on fetal hormonal and hemodynamic stress response to intrauterine needling. Anesthesiology. 2001 Oct;95(4):828-35. doi: 10.1097/00000542-200110000-00008. PMID 11605920
- [Result] Cauldwell CB. Anesthesia for fetal surgery. Anesthesiol Clin North Am. 2002 Mar;20(1):211-26. doi: 10.1016/s0889-8537(03)00062-2. PMID 11892506
- [Result] Devoto JC, Alcalde JL, Otayza F, Sepulveda W. Anesthesia for myelomeningocele surgery in fetus. Childs Nerv Syst. 2017 Jul;33(7):1169-1175. doi: 10.1007/s00381-017-3437-7. Epub 2017 May 25. PMID 28547209